CLINICAL TRIAL: NCT00005346
Title: Mechanisms Underlying Abnormal Ambulatory BP Patterns
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4215; R01HL046177 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2001-11

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

SUMMARY:
To understand the mechanism(s) underlying sodium-dependent blood pressure control, and to determine the consequences thereof.

DETAILED DESCRIPTION:
BACKGROUND:

The blood pressure of a significant percentage of the hypertensive population, and the normotensive population at a high risk for the development of hypertension (Blacks and older individuals), is sodium (salt)-dependent. That is to say, increasing the intake of salt will increase blood pressure in these individuals; conversely, and more importantly, decreasing the intake of salt will reduce blood pressure.

DESIGN NARRATIVE:

The investigators believed that the mechanisms responsible for sodium-dependent blood pressure were only indirectly linked to race, sex, and age. Their research was consistent with the hypothesis that sodium-dependent blood pressure control resulted from decreased responsiveness of the renal and adrenal blood pressure regulatory systems. This produced abnormal daily blood pressure patterns, with reduced fluctuation resulting in extended periods of increased blood pressure. The increased cardiovascular load led to the early development of cardiovascular and renal disease, including hypertension. They tested this hypothesis by identifying 'high risk' and 'normal risk' subjects based on renal responses to sodium restriction. The subjects were equal numbers of healthy males and females, Blacks and whites, between the ages of 55-70 years. Using an innovative approach, they then examined the influence of risk status on 24-hour patterns of blood pressure, hormonal activity, and sodium handling. Finally, they determined the clinical significance of the profiles by examining changes in cardiac and renal status at a two-year follow-up.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1993-01; Study Completion 1995-12 (Actual)